CLINICAL TRIAL: NCT00003336
Title: A Pilot Study of Unrelated Umbilical Cord Blood Transplantation in Patients With Severe Aplastic Anemia, Inborn Errors in Metabolism, or Inherited Hematologic Stem Cell Disorders
Brief Title: Pilot Study Of Unrelated UCB Transplant for Non-Malignant Hematologic Conditions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Mary J. Laughlin, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU5Y97; P30CA043703 (NIH); CASE-CWRU-5Y97; NCI-G98-1431; CASE-5Y97
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Anemia, Refractory; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Melphalan; Methylprednisolone; Cord Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin — The regimen varies according to the underlying cause of the anemia.Patients receive high-dose chemotherapy and/or radiotherapy as a conditioning regimen beginning 6-9 days before the umbilical cord blood transplant (UCBT).
Drug: busulfan — The regimen varies according to the underlying cause of the anemia.Patients receive high-dose chemotherapy and/or radiotherapy as a conditioning regimen beginning 6-9 days before the umbilical cord blood transplant (UCBT).
Drug: cyclophosphamide — The regimen varies according to the underlying cause of the anemia.Patients receive high-dose chemotherapy and/or radiotherapy as a conditioning regimen beginning 6-9 days before the umbilical cord blood transplant (UCBT).
Drug: melphalan — The regimen varies according to the underlying cause of the anemia.Patients receive high-dose chemotherapy and/or radiotherapy as a conditioning regimen beginning 6-9 days before the umbilical cord blood transplant (UCBT).
Drug: methylprednisolone — The regimen varies according to the underlying cause of the anemia.Patients receive high-dose chemotherapy and/or radiotherapy as a conditioning regimen beginning 6-9 days before the umbilical cord blood transplant (UCBT).
Procedure: bone marrow ablation with stem cell support
Procedure: umbilical cord blood transplantation — One day after the conditioning regimen is completed, patients receive the UCBT.
Radiation: radiation therapy — The regimen varies according to the underlying cause of the anemia.Patients receive high-dose chemotherapy and/or radiotherapy as a conditioning regimen beginning 6-9 days before the umbilical cord blood transplant (UCBT).

SUMMARY:
RATIONALE: Umbilical cord blood transplantation may allow doctors to give higher doses of chemotherapy or radiation therapy and kill more cancer cells.

PURPOSE: This phase II trial is studying how well umbilical cord blood transplantation works in treating patients with severe aplastic anemia, malignant thymoma, or myelodysplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the rates of durable engraftment in patients with severe aplastic anemia, myelodysplastic syndrome, inborn errors of metabolism, or inherited hematopoietic disorders, refractory to medical management, who are undergoing high-dose chemoradiotherapy followed by unrelated cord blood (UCB) transplantation.
* Evaluate the rate and quality of immunologic reconstitution in this patient population.

OUTLINE: Patients are stratified according to weight (under 45 kg vs over 45 kg).

Patients receive high-dose chemotherapy and/or radiotherapy as a conditioning regimen beginning 6-9 days before the umbilical cord blood transplant (UCBT). The regimen varies according to the underlying cause of the anemia, but could include busulfan, cyclophosphamide or melphalan, anti-thymocyte globulin or methylprednisolone, and/or radiation therapy. One day after the conditioning regimen is completed, patients receive the UCBT.

Patients are followed weekly for 3 months, at 6 months, then every 6 months for 2.5 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 4-90 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of severe aplastic anemia based on bone marrow cellularity of less than 20%
* Must meet at least two of the following criteria:

  * Granulocyte count less than 500/mm^3
  * Platelet count less than 20,000/mm^3
  * Reticulocyte count less than 50,000/mm^3
* Following etiologies eligible:

  * Fanconi's anemia
  * Hypoplastic leukemia
  * Monosomy 7
  * Drug exposure (chloramphenicol, NSAIDS)
  * Viral exposure (EBV, hepatitis, parvovirus, HIV)
  * Nutritional deficiencies
  * Thymoma
  * Paroxysmal nocturnal hemoglobinuria
  * Amegakaryocytic thrombocytopenia OR
* Histologically confirmed myelodysplastic syndrome (MDS) that is refractory to medical management or with cytogenic abnormalities predictive of transformation into acute leukemia, including 5q-, 7q-, monosomy 7, or trisomy 8
* The following etiologies only are eligible:

  * Refractory anemia
  * Refractory anemia with ringed sideroblasts
  * De novo primary MDS
  * Therapy-related secondary MDS OR
* Confirmed diagnosis of inherited hematopoietic disorder that is refractory to medical management
* Following etiologies eligible:

  * Severe combined immunodeficiency
  * Familial erythrophagocytic lymphohistiocytosis
  * Wiskott-Aldrich syndrome
  * Kostmann's syndrome (infantile histiocytosis)
  * Chronic granulomatous disease
  * Leukocytic adhesion deficiency
  * Chediak-Higashi syndrome
  * Paroxysmal nocturnal hemoglobinuria
  * Fanconi's anemia
  * Dyskeratosis congenita
  * Diamond-Blackfan anemia
  * Amegakaryocytic thrombocytopenia
  * Osteopetrosis
  * Gaucher's disease
  * Lesch-Nyhan syndrome
  * Mucopolysaccharidoses
  * Lipodoses
* Autologous or haploidentical related peripheral blood stem cells available as backup
* Serologically matched umbilical cord blood unit available in the New York Blood Center's Placental Blood Project, or other acceptable umbilical cord blood registry

PATIENT CHARACTERISTICS:

Age:

* 55 and under

Performance status:

* Zubrod 0-1
* Karnofsky 80-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* See Disease Characteristics

Hepatic:

* ALT/AST no greater than 4 times normal
* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 2.0 mg/dL
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* Normal cardiac function by echocardiogram or radionuclide scan
* Shortening fraction or ejection fraction at least 80% normal for age
* Non-Fanconi patients with acquired or congenital cardiomyopathy may receive melphalan as a substitute for cyclophosphamide

Pulmonary:

* FVC and FEV_1 at least 60% of predicted for age
* DLCO at least 60% of predicted in adult patients

Other:

* No active concurrent malignancy
* No active infection
* Not pregnant or nursing
* HIV negative
* Must have an available serologic matched Umbilical Cord Blood Unit (UCBU) in the New York Blood Center's Placental Blood Project, or other acceptable Umbilical Cord Blood (UCB) registry

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No concurrent cytotoxic chemotherapy

Endocrine therapy:

* No concurrent immunosuppressive medications

Radiotherapy:

* No concurrent radiotherapy

Surgery:

* Not specified

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 1998-01; Primary Completion 2005-12 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Event-free survival by disease assessment | at 100 days and at 6, 9, 12, 18, and 24 months

SECONDARY OUTCOMES:
Umbilical cord blood donor engraftment by chimerism and complete blood count (CBC) at time of myeloid recovery. | 100 days and at 6, 9, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary J. Laughlin, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Laughlin MJ, Barker J, Bambach B, Koc ON, Rizzieri DA, Wagner JE, Gerson SL, Lazarus HM, Cairo M, Stevens CE, Rubinstein P, Kurtzberg J. Hematopoietic engraftment and survival in adult recipients of umbilical-cord blood from unrelated donors. N Engl J Med. 2001 Jun 14;344(24):1815-22. doi: 10.1056/NEJM200106143442402. PMID 11407342